Study Title: PrEPARE: PrEP in Pregnancy, Accelerating Reach and Efficiency

**NCT#**: 04712994

Principal Investigator: Grace John-Stewart, MD, PhD, MPH

**Document Name:** Oral Consent Guide

**IRB Approval Date:** December 17, 2020

#### **Oral Consent Guide**

| NAME | POSITION | DEPARTMENT | TELEPHONE<br>NUMBERS |
|---|---|---|---|
| Grace John-Stewart | Co-Principal Investigator | Global Health, UW | +1-206-543-4278 |
| Pamela Kohler | Co-Principal Investigator | Psychosocial &<br>Community Health, UW | +1-206-616-7962 |
| Anjuli Wagner | Co-Principal Investigator | Global Health, UW | +1-978-460-2331 |
| John Kinuthia | Site Principal Investigator | Kenyatta National<br>Hospital | +254-0722-799-052 |
| Felix Abuna | Assistant Coordinator | Kenyatta National<br>Hospital | +254721230652 |
| Nancy Mwongeli | Study Coordinator | Kenyatta National<br>Hospital | +254713 917 226 |

Emergency telephone number: John Kinuthia +254 0722 799 052

# It is important to cover the following topics with the study participants: Background information:

- Kenyatta National Hospital and the University of Washington are conducting a study to determine the best way to provide PrEP to women in MCH and FP clinics.
- Goal is to identify the best way to reach women who are in need or may benefit from PrEP as an HIV prevention strategy.

### Benefits of program:

The program will help learn the best ways to deliver PrEP to women who need it in Kenya.

#### Procedures:

Time and Motion

Participants may also be asked to carry a form for providers to note the start and end time of each service they
receive.

#### Exit Survey

We will ask questions about knowledge of PrEP and experiences at the clinic.

## The risks and discomfort related to this program:

- Participants may may feel uncomfortable answering some of the questions today. There are no correct answers and we want to know their thoughts an opinions.
- All efforts shall be made to keep information private and confidential. We will not collect or record participant names today to help keep responses private.

#### **Benefits:Compensation**

• There is no compensation for participation

## Confidentiality of Research Information

The information provided will be kept secret by the study staff. We will not publish or discuss in public anything that could identify participants.

#### Other information:

- A description of this clinical trial will be available on <a href="http://www.clinicaltrials.gov">http://www.clinicaltrials.gov</a>, as required by US Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.
- participation in this study is voluntary.
- Participants do not have to be in this study if they do not want to,
- Answer any questions they may have and give them clinic contact information for future questions.

#### Final Step:

- Ensure the participant understands what the survey is about and if they have any questions
- After you answer their questions verbally confirm that they agree to participant in the survey today.

# All participants:

□ Confirm the participant is willing to participate, remind them they are not forced to participate in any activities and may chose not to answer any question at any time.

PrEPARE Exit Survey Oral Consent Guide v1.2

